CLINICAL TRIAL: NCT04700137
Title: Investigating the Mental Health Impact of COVID-19 and Comparing the Effectiveness of Two Caring Contact Interventions on Patients, Providers, and Staff of St. Luke's Health System
Brief Title: Mental Health Among Patients, Providers, and Staff During the COVID-19 Era
Acronym: MHAPPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's Health System, Boise, Idaho (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Idaho Crisis & Suicide Hotline (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Anna Radin, Applied Research Scientist, St. Luke's Health System, Boise, Idaho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-0052; PCORI HIS-2018C3-14695 (Other Grant/Funding Number: COVID-19 Enhancement Award, PCORI)
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Results first posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-05

CONDITIONS: Covid19; Mental Health
Keywords: Loneliness; Anxiety; Depression; Suicidal Ideation; Social Distancing; Mental Distress; Pandemic; Caring Contacts; Healthcare Staff; Healthcare Providers; Brief Contact Intervention; Adults; Adolescents
MeSH Terms: conditions — COVID-19; Psychological Well-Being; Anxiety Disorders; Depression; Suicidal Ideation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caring Contacts + Introductory Phone Call (CC+) (Active Comparator): Healthcare provider and staff participants who are randomized to both caring text messages and an introductory phone call.
  Adult and adolescent participants who are randomized to both caring text messages and an introductory phone call.
  Interventions: Other: Caring Contacts Plus Introductory Phone Call (CC+)
- Caring Contacts (without phone call) (CC) (Active Comparator): Healthcare provider and staff participants who are randomized to only caring text messages.
  Adult and adolescent patient participants who are randomized to only caring text messages.
  Interventions: Other: Caring Contacts without an introductory phone call (CC)

INTERVENTIONS:
Other: Caring Contacts Plus Introductory Phone Call (CC+) — One introductory semi-structured caring phone conversation with a follow-up specialist to check-in, establish a personal connection, and provide resources at the 0-2 week time-point followed by 11 non-demanding, caring text or email messages sent over the course of 6 months.
  Arms: Caring Contacts + Introductory Phone Call (CC+)
Other: Caring Contacts without an introductory phone call (CC) — Eleven non-demanding, caring text or email messages sent over the course of 6 months. Participants will not know or have spoken to the follow-up specialist who sends the caring messages.
  Arms: Caring Contacts (without phone call) (CC)

SUMMARY:
The Mental Health Among Patients, Providers, and Staff (MHAPPS) Study is designed to study how the COVID-19 pandemic has affected mental health and wellbeing, and how to support mental health while minimizing the burden on the healthcare system. The study will enroll adults and adolescents who have had a primary care visit in the last 12 months, as well as healthcare providers and staff from a large health system in Idaho.

The study will include:

Aim 1: a cross sectional survey to measure the prevalence of various measures of mental distress and how they are associated with COVID-19-related factors; and

Aim 2: a randomized controlled trial comparing the effectiveness of two versions of a Caring Contacts intervention to reduce loneliness and mental distress.

DETAILED DESCRIPTION:
Approximately 4,800 participants will complete the Aim 1 survey. The Caring Contacts intervention involves sending a series of brief, non-demanding, supportive text messages to the participant. One intervention arm will receive an introductory phone call and the caring text messages (CC+); the second intervention arm will only receive the same caring text messages (CC). The clinical trial will enroll a subset of 660 participants who report elevated levels of loneliness, suicide ideation, or other mental distress in the Aim 1 survey. Enrollment will be stratified by population (providers and employees; patients) with 165 per intervention arm in each stratum.

The investigators hypothesize that delivering the Caring Contacts intervention with an introductory phone call will yield better mental health outcomes than delivering the Caring Contacts intervention with no introductory phone call.

This will be the first published data directly comparing the effectiveness of two versions of the Caring Contacts intervention with individuals who report loneliness or other mental distress. The overall goal of the MHAPPS study is to better understand the mental health impact of COVID-19 and to determine how health systems can most effectively support mental health at scale among providers, staff, and patients in the COVID-19 era and beyond.

This research is being conducted by a team including health system-based researchers, clinicians, other frontline healthcare workers, and administrators; academic researchers; follow-up specialists and administrators at the Idaho Suicide Prevention Hotline, and an advisory board of people with lived experience with suicide.

ELIGIBILITY:
Inclusion Criteria:

Aim 1:

* Provider & Employee Inclusion Criteria

  * Provider or Employee at St. Luke's Health System
  * Adults ≥ 18 years of age
  * Proficient in spoken and written English language
* Patient Inclusion Criteria

  * Patient at a St. Luke's Health System primary care site
  * Current MyChart account user
  * Adults ≥18 years of age
  * Minors 12-17 years of age
  * Proficient in spoken and written English language

Aim 2:

* Provider & Employee Inclusion Criteria

  * Moderate or high score for loneliness, suicide ideation, psychological stress, anxiety, or depression:

    * NIH Toolkit Loneliness raw score of 13 or greater or
    * C-SSRS score of 3 or greater; or
    * NIH Toolkit Perceived Stress raw score of 31 or greater for adults; or
    * GAD7 score of 11 or greater; or
    * PHQ9 score of 10 or greater
  * Access to a phone for the duration of the study with the ability to receive text messages and phone calls
* Patient Inclusion Criteria

  * Moderate or high score for loneliness, suicide ideation, psychological stress, anxiety, or depression:

    * NIH Toolkit Loneliness raw score of 13 or greater for adults or 16 or greater for adolescents; or
    * C-SSRS score of 3 or greater; or
    * GAD7 score of 11 or greater; or
    * PHQ9 score of 10 or greater; or
    * NIH Toolkit Stress raw score of 31 or greater for adults or 33 or greater for adolescents
    * [Note: validated youth versions of the NIH Toolkit assessments (loneliness and perceived stress), and PHQ-A tools will be used for adolescents; the C-SSRS and GAD7 tools are validated for use with both adults and adolescents.]
  * Access to a phone for the duration of the study with the ability to receive text messages and phone calls

Exclusion Criteria:

Aim 1:

* Provider & Employee Exclusion Criteria

  * Individuals who are unable or unwilling to provide informed consent to participate
  * Individuals who are study staff for this study or the SPARC Trial
* Patient Exclusion Criteria

  * Individuals who are unable or unwilling to provide informed consent to participate.
  * Individuals who are participants in the SPARC Trial
  * Individuals who have not had a primary care visit in the past 12 months

Aim 2:

* Provider & Employee Exclusion Criteria

  * Individuals who are unable or unwilling to provide informed consent to participate
  * Individuals who are in acute crisis as determined by the person conducting the consent process
  * Individuals who are study staff for this study or the SPARC Trial
  * Individuals who are enrolled as participants in the SPARC comparative effectiveness clinical trial (SPARC Aim 1). Providers or employees who received training related to SPARC and/or who completed the SPARC provider satisfaction survey are not excluded from participating in MHAPPS
* Patient Exclusion Criteria

  * Patients who are unable or unwilling to provide informed consent/assent to participate (or whose legally authorized representative is unable or unwilling to provide consent in the case of adolescents). Examples may include but are not limited to patients who present with acute or chronic cognitive impairment that would preclude their ability to consent (i.e. acute psychosis, intoxication, or intellectual disability).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 666 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna K Radin, DrPH, MPH, Principal Investigator — St. Luke's Health System
Locations (1):
- St. Luke's Health System, Boise, Idaho, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested from other researchers 5 years after the completion of the primary endpoint by contacting the PIs.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 5 years following the completion of the primary endpoint
Access Criteria: Data from this trial may be requested by other researchers 5 years after the completion of the primary endpoint by contacting the PI. The PI will ensure all mechanisms used to share data will include proper plans and safeguards for the protection of privacy, confidentiality, and security for data dissemination and reuse (e.g., all data will be thoroughly de-identified and will not be traceable to a specific study participant).

REFERENCES:
- [Derived] Radin AK, Shaw J, Brown SP, Torres J, Harper M, Flint H, Fouts T, McCue E, Skeie A, Pena C, Youell J, Doty-Jones A, Wilson J, Flinn L, Austin G, Chan KCG, Zheng Z, Fruhbauerova M, Walton M, Kerbrat A, Comtois KA. Comparative effectiveness of two versions of a caring contacts intervention in healthcare providers, staff, and patients for reducing loneliness and mental distress: A randomized controlled trial. J Affect Disord. 2023 Jun 15;331:442-451. doi: 10.1016/j.jad.2023.03.029. Epub 2023 Mar 22. PMID 36963515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between January 2021 and July 2021. All recruitment was completed virtually, with invitations to participate sent via email and via the electronic health record messaging service.
Pre-assignment Details: Randomization occurred once a potential participant joined a study enrollment phone call but before they consented to participate. This approach was practical given the electronic nature of the informed consent process and was recommended by the Data & Safety Monitoring Committee as a way to include a description in writing of the assigned intervention on the informed consent form while masking participants to the details of the intervention arm to which they were not assigned.
Groups:
- Patients -- Caring Contacts (Without Phone Call) (CC): Patients randomized to only caring text messages.
  Caring Contacts without an introductory phone call (CC): Eleven non-demanding, caring text or email messages sent over the course of 6 months. Participants will not know or have spoken to the follow-up specialist who sends the caring messages.
- Patients -- Caring Contacts + Introductory Phone Call (CC+): Patients randomized to caring text messages and an introductory phone call.
  Caring Contacts Plus Introductory Phone Call (CC+): One introductory semi-structured caring phone conversation with a follow-up specialist to check-in, establish a personal connection, and provide resources at the 0-2 week time-point followed by 11 non-demanding, caring text or email messages sent over the course of 6 months.
- Healthcare Providers/Staff -- Caring Contacts (Without Phone Call) (CC): Healthcare Providers and staff randomized to only caring text messages.
  Caring Contacts without an introductory phone call (CC): Eleven non-demanding, caring text or email messages sent over the course of 6 months. Participants will not know or have spoken to the follow-up specialist who sends the caring messages.
- Healthcare Providers/Staff -- Caring Contacts + Introductory Phone Call (CC+): Healthcare providers and staff randomized to caring text messages and an introductory phone call.
  Caring Contacts Plus Introductory Phone Call (CC+): One introductory semi-structured caring phone conversation with a follow-up specialist to check-in, establish a personal connection, and provide resources at the 0-2 week time-point followed by 11 non-demanding, caring text or email messages sent over the course of 6 months.
Period: Overall Study
Arm/Group | Patients -- Caring Contacts (Without Phone Call) (CC) | Patients -- Caring Contacts + Introductory Phone Call (CC+) | Healthcare Providers/Staff -- Caring Contacts (Without Phone Call) (CC) | Healthcare Providers/Staff -- Caring Contacts + Introductory Phone Call (CC+)
Started (Randomized and consented.) | 166 | 165 | 168 | 167
Completed (Completed the study, including the entire final outcome survey.) | 165 | 159 | 165 | 166
Not Completed | 1 | 6 | 3 | 1
Not completed — Lost to Follow-up | 1 | 6 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients - CC: Patients randomized to Caring Contacts without an introductory phone call (CC) intervention arm
- Patients - CC+: Patients randomized to Caring Contacts with an introductory phone call (CC+) intervention arm
- Healthcare Providers/Staff - CC: Healthcare providers and staff randomized to Caring Contacts without an introductory phone call (CC) intervention arm
- Healthcare Providers/Staff - CC+: Healthcare providers and staff randomized to Caring Contacts with an introductory phone call (CC+) intervention arm
- Total: Total of all reporting groups
Arm/Group | Patients - CC | Patients - CC+ | Healthcare Providers/Staff - CC | Healthcare Providers/Staff - CC+ | Total
Number analyzed (Participants) | 166 | 165 | 168 | 167 | 666
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (17) | 47.2 (15.8) | 42.1 (12.2) | 40.6 (11.3) | 43.1 (14.4)
Age, Continuous [Median (Full Range); unit: years] | 43.8 [12.9 to 89.4] | 46.6 [18 to 83.9] | 39.8 [20.5 to 69.6] | 39.5 [22 to 72.2] | 41 [12.9 to 89.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 131 | 140 | 150 | 551
  Male | 36 | 34 | 28 | 17 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 12 | 19 | 51
  Not Hispanic or Latino | 156 | 154 | 153 | 145 | 608
  Unknown or Not Reported | 1 | 0 | 3 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 2
  Asian | 3 | 1 | 1 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 2
  Black or African American | 2 | 1 | 1 | 0 | 4
  White | 153 | 156 | 155 | 157 | 621
  More than one race | 4 | 4 | 7 | 5 | 20
  Unknown or Not Reported | 1 | 3 | 3 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 166 | 165 | 168 | 167 | 666
Health System Employee Type [Count of Participants; unit: Participants] — Population: Health system employee type was only assessed for healthcare providers and staff.
  Participants
    Physicians & Advanced Practice Providers: number analyzed (Participants) | 0 | 0 | 168 | 167 | 335
    Physicians & Advanced Practice Providers |  |  | 8 | 8 | 16
    Pharmacy, Patient Access Specialists, Lab: number analyzed (Participants) | 0 | 0 | 168 | 167 | 335
    Pharmacy, Patient Access Specialists, Lab |  |  | 26 | 20 | 46
    Trades & Food Service: number analyzed (Participants) | 0 | 0 | 168 | 167 | 335
    Trades & Food Service |  |  | 1 | 2 | 3
    Nursing: number analyzed (Participants) | 0 | 0 | 168 | 167 | 335
    Nursing |  |  | 57 | 67 | 124
    Office Work & Educators: number analyzed (Participants) | 0 | 0 | 168 | 167 | 335
    Office Work & Educators |  |  | 62 | 60 | 122
    Senior Management: number analyzed (Participants) | 0 | 0 | 168 | 167 | 335
    Senior Management |  |  | 2 | 2 | 4
    Social Support Services: number analyzed (Participants) | 0 | 0 | 168 | 167 | 335
    Social Support Services |  |  | 11 | 6 | 17
    Other: number analyzed (Participants) | 0 | 0 | 168 | 167 | 335
    Other |  |  | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Loneliness as Measured by the National Institutes of Health (NIH) Toolbox Social Relationship Scale for Loneliness
Description: The NIH Toolbox Social Relationship Scale for Loneliness is a validated method for measuring loneliness. Participants rate items on a 5-point scale, with options ranging from never (1) to always (5). This creates a raw score, which is then converted to a t-score, with higher scores indicating greater levels of loneliness. T-score of 50 represents the mean of the US general population (based on the 2010 Census) and 10 T-score units represents one standard deviation. A T-score of 60.7 or more (adults) or 60 or more (youth) indicates moderate to high levels of loneliness.
Time Frame: Baseline and 6 Months
Population: Intention to treat population - all participants who were randomized and consented.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Patients - CC | Patients - CC+ | Healthcare Providers/Staff - CC | Healthcare Providers/Staff - CC+
Number analyzed (Participants) | 166 | 165 | 168 | 167
T-score
  Baseline Loneliness | 64.4 (9.9) | 64.4 (10.3) | 62.6 (9.3) | 62.5 (9.5)
  Follow-up Loneliness (6 months) | 61.9 (10.7) | 60.8 (10.3) | 61.2 (11) | 61.3 (11.1)
Statistical Analysis 1: Comparison: Patients - CC vs Patients - CC+; Difference in loneliness among patients by intervention arm at follow-up (6 months); Test type: Superiority; p = 0.31, Regression, Linear — p<0.05 = a priori threshold for statistical significance; Linear regression with robust standard errors, adjusting for the baseline score as a precision variable; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-3.0 to 1.0] — A T-score of 50 represents the mean of the US general population (based on the 2010 Census) and 10 T-score units represents one standard deviation. Higher T-score indicates higher loneliness
Statistical Analysis 2: Comparison: Healthcare Providers/Staff - CC vs Healthcare Providers/Staff - CC+; Difference in loneliness among healthcare providers/staff by intervention arm at follow-up (6 months); Test type: Superiority; p = 0.83, Regression, Linear — p<0.05 = a priori threshold for statistical significance; Linear regression with robust standard errors, adjusting for the baseline score as a precision variable; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.8 to 2.2] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Suicidal Ideation & Behavior as Measured by the Columbia Suicide Severity Rating Scale
Description: The Columbia Suicide Severity Rating Scale (C-SSRS) 6-item screener (self-assessment lifetime-recent (baseline) and since last visit (6 months) for Primary Care settings versions will be used). The C-SSRS is a validated tool to assess suicidality. C-SSRS score is determined based on the highest question number to which the participant responds "yes". For example, a score of 5 would be assigned to a participant who responded "yes" to Question 5 and any or all preceding questions. Higher scores are indicative of greater risk for suicide. C-SSRS screener scores range from 0 to 6, with higher scores indicative of higher suicide risk. Scores of 3 and higher indicate moderate to high risk for suicide.
Time Frame: Baseline and 6 Months
Population: The Intention to Treat population includes data for all participants who were randomized, completed study enrollment, and completed the baseline survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients - CC | Patients - CC+ | Healthcare Providers/Staff - CC | Healthcare Providers/Staff - CC+
Number analyzed (Participants) | 166 | 165 | 168 | 167
score on a scale
  Baseline C-SSRS | 0.5 (1.3) | 0.4 (1.1) | 0.3 (0.9) | 0.4 (1.1)
  Follow-up C-SSRS (6 months) | 0.4 (0.9) | 0.6 (1.3) | 0.5 (1.2) | 0.4 (1.1)
Statistical Analysis 1: Comparison: Patients - CC vs Patients - CC+; Difference in suicidal ideation and behavior (C-SSRS) among patients by intervention arm at follow-up (6 months); Test type: Superiority; p = 0.05, Regression, Linear — p<0.05 = a priori threshold for statistical significance; Linear regression with robust standard errors, adjusting for the baseline score as a precision variable; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [0.0 to 0.5]
Statistical Analysis 2: Comparison: Healthcare Providers/Staff - CC vs Healthcare Providers/Staff - CC+; Difference in suicidal ideation and behavior (C-SSRS) among healthcare providers/staff by intervention arm at follow-up (6 months); Test type: Superiority; p = 0.2, Regression, Linear — p<0.05 = a priori threshold for statistical significance; Linear regression with robust standard errors, adjusting for the baseline score as a precision variable; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.1]

3. Secondary Outcome: Depression as Measured by the Patient Health Questionnaire (PHQ-9)
Description: The PHQ-9 is a widely used and validated tool to screen for depression in primary care and other non-psychiatric settings. The tool is composed of 9 questions each with a response of 0-3 which generate a score from 0-27 with higher scores indicating a greater degree of depression. Scores are categorized in the following manner: a score of 5-9 is considered minimal depression, 10-14 is considered mild major, 15-19 is moderate major, and ≥20 is severe major.
Time Frame: Baseline and 6 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients - CC | Patients - CC+ | Healthcare Providers/Staff - CC | Healthcare Providers/Staff - CC+
Number analyzed (Participants) | 166 | 165 | 168 | 167
score on a scale
  Baseline PHQ-9 | 10.5 (6.1) | 10.0 (6.0) | 8.4 (5.0) | 8.6 (5.4)
  Follow-up PHQ-9 (6 months) | 8.6 (6.2) | 7.9 (5.8) | 7.7 (5.1) | 8.1 (5.4)
Statistical Analysis 1: Comparison: Patients - CC vs Patients - CC+; Difference in depression (PHQ-9) among patients by intervention arm at follow-up (6 months); Test type: Superiority; p = 0.45, Regression, Linear — p<0.05 = a priori threshold for statistical significance; Linear regression with robust standard errors, adjusting for the baseline score as a precision variable; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.5 to 0.7]
Statistical Analysis 2: Comparison: Healthcare Providers/Staff - CC vs Healthcare Providers/Staff - CC+; Difference in depression (PHQ-9) among healthcare providers/staff by intervention arm at follow-up (6 months); Test type: Superiority; p = 0.51, Regression, Linear — p<0.05 = a priori threshold for statistical significance; Linear regression with robust standard errors, adjusting for the baseline score as a precision variable; Median Difference (Final Values) = 0.3, 95% CI 2-sided [-0.7 to 1.3]

4. Secondary Outcome: Anxiety as Measured by the Generalized Anxiety Disorder 7 Item Scale (GAD-7)
Description: Symptoms of anxiety will be assessed using the GAD-7, a brief self-report scale frequently used in the identification of Generalized Anxiety Disorder. The tool is composed of seven items, which are rated 0-3 to generate a score from 0-21. Higher scores indicate a greater severity of generalized anxiety symptoms. Scores of 11 and higher indicate moderate to high anxiety.
Time Frame: Baseline and 6 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients - CC | Patients - CC+ | Healthcare Providers/Staff - CC | Healthcare Providers/Staff - CC+
Number analyzed (Participants) | 166 | 165 | 168 | 167
score on a scale
  Baseline GAD-7 | 9.3 (5.3) | 8.8 (5.3) | 7.8 (4.4) | 8.4 (5.0)
  Follow-up GAD-7 (6 months): number analyzed (Participants) | 165 | 159 | 165 | 166
  Follow-up GAD-7 (6 months) | 7.9 (5.6) | 7.3 (5.0) | 6.8 (4.7) | 8.2 (5.1)
Statistical Analysis 1: Comparison: Patients - CC vs Patients - CC+; Difference in anxiety (GAD-7) among patients by intervention arm at follow-up (6 months); Test type: Superiority; p = 0.54, Regression, Linear — p<0.05 = a priori threshold for statistical significance; Linear regression with robust standard errors, adjusting for the baseline score as a precision variable; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.3 to 0.7]
Statistical Analysis 2: Comparison: Healthcare Providers/Staff - CC vs Healthcare Providers/Staff - CC+; Difference in anxiety (GAD-7) among healthcare providers/staff by intervention arm at follow-up (6 months); Test type: Superiority; p = 0.04, Regression, Linear — p<0.05 = a priori threshold for statistical significance; Linear regression with robust standard errors, adjusting for the baseline score as a precision variable; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [0.1 to 2.0]

5. Secondary Outcome: Change From Baseline in Psychological Stress as Measured by the National Institutes of Health (NIH) Toolbox Stress and Self-Efficacy Scales Perceived Stress Measure
Description: The National Institute of Health (NIH) Toolbox Self-Efficacy Scales Perceived Stress measure is a validated tool to measure the stress and coping resources of an individual. The measure is comprised of ten items which are scored and granted a t-score specific to adult or adolescent participants. Higher t-scores are indicative of higher levels of stress. T-score of 50 represents the mean of the US general population (based on the 2010 Census) and 10 T-score units represents one standard deviation. A T-score of 60.5 or more for adults or 60.8 or more in adolescents indicates moderate to high levels of stress.
Time Frame: Baseline and 6 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Patients - CC | Patients - CC+ | Healthcare Providers/Staff - CC | Healthcare Providers/Staff - CC+
Number analyzed (Participants) | 166 | 165 | 168 | 167
T-score
  Baseline Perceived Stress | 60.7 (8.7) | 59.6 (8.6) | 58.5 (7.3) | 59.5 (7.7)
  Follow-up Perceived Stress (6 months): number analyzed (Participants) | 165 | 159 | 165 | 166
  Follow-up Perceived Stress (6 months) | 56.5 (10.7) | 55.3 (10.1) | 55.1 (9.2) | 57.6 (9.6)
  Change in Perceived Stress from Baseline to 6 months: number analyzed (Participants) | 165 | 159 | 165 | 166
  Change in Perceived Stress from Baseline to 6 months | -4.2 (9.3) | -4.4 (8.0) | -3.3 (10.3) | -1.9 (9.9)
Statistical Analysis 1: Comparison: Patients - CC vs Patients - CC+; Change in stress from baseline to 6 months among patients; Test type: Superiority; p = 0.84, Regression, Linear — p<0.05 = a priori threshold for statistical significance; Linear regression with robust standard errors; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.1 to 1.7] — T-score of 50 = mean of the US general population (2010 Census); 10 T-score units = one standard deviation. Higher T-scores = higher stress. T-scores equal to or greater than 60.5 (adults) or 60.8 (adolescents) are moderate or high risk
Statistical Analysis 2: Comparison: Healthcare Providers/Staff - CC vs Healthcare Providers/Staff - CC+; Change in stress from baseline to 6 months among healthcare providers/staff; Test type: Superiority; p = 0.18, Regression, Linear — p<0.05 = a priori threshold for statistical significance; Linear regression with robust standard errors; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-0.7 to 3.7] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Perceived Burdensomeness & Thwarted Belongingness as Measured by the Interpersonal Needs Questionnaire (INQ15)
Description: The Interpersonal Needs Questionnaire (INQ) was developed from the Interpersonal Theory of Suicide and the 15-item version (INQ15) is a validated tool to measure both perceived burdensomeness (PB) (6 items, scores range from 6 to 42) and thwarted belongingness (TB) (9 items; scores range from 9 to 63). Individuals provide a self-report response to each item ranging from 1 (Not at all true for me) to 7 (Very true for me). The appropriate items are reverse coded, and items are summed to calculate the TB and PB subscale scores with higher scores indicating greater TB and PB. Clinical Cutoff scores predicting desire for death are 35 or greater for TB and 19 or greater for PB. Clinical cutoff scores predicting desire for suicide are 50 or greater for TB and 30 or greater for PB.
Time Frame: Baseline and 6 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients - CC | Patients - CC+ | Healthcare Providers/Staff - CC | Healthcare Providers/Staff - CC+
Number analyzed (Participants) | 166 | 165 | 168 | 167
score on a scale
  Baseline INQ Perceived Burdensomeness | 10.1 (6.7) | 9.2 (5.4) | 7.9 (3.6) | 8.0 (4.9)
  Follow-up INQ Perceived Burdensomeness (6 months) | 9.6 (6.8) | 9.5 (6.7) | 8.4 (5.1) | 8.5 (5.1)
  Baseline INQ Thwarted Belongingness | 31.1 (11.1) | 30.3 (11.4) | 31.4 (10.0) | 30.4 (11.8)
  Follow-up INQ Thwarted Belongingness (6 months) | 29.3 (12.2) | 27.6 (12.3) | 27.8 (12.3) | 28.6 (12.4)
Statistical Analysis 1: Comparison: Patients - CC vs Patients - CC+; Difference in perceived burdensomeness (INQ15) among patients by intervention arm at follow-up (6 months); Test type: Superiority; p = 0.38, Regression, Linear — p<0.05 = a priori threshold for statistical significance; Linear regression with robust standard errors, adjusting for the baseline score as a precision variable; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.6 to 1.6]
Statistical Analysis 2: Comparison: Healthcare Providers/Staff - CC vs Healthcare Providers/Staff - CC+; Difference in perceived burdensomeness (INQ15) among healthcare providers/staff by intervention arm at follow-up (6 months); Test type: Superiority; p = 0.81, Regression, Linear — p<0.05 = a priori threshold for statistical significance; Linear regression with robust standard errors, adjusting for the baseline score as a precision variable; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.8 to 1.0]
Statistical Analysis 3: Comparison: Patients - CC vs Patients - CC+; Difference in thwarted belongingness (INQ15) among patients by intervention arm at follow-up (6 months); Test type: Superiority; p = 0.73, Regression, Linear — p<0.05 = a priori threshold for statistical significance; Linear regression with robust standard errors, adjusting for the baseline score as a precision variable; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.6 to 1.8]
Statistical Analysis 4: Comparison: Healthcare Providers/Staff - CC vs Healthcare Providers/Staff - CC+; Difference in thwarted belongingness (INQ15) among healthcare providers/staff by intervention arm at follow-up (6 months); Test type: Superiority; p = 0.24, Regression, Linear — p<0.05 = a priori threshold for statistical significance; Linear regression with robust standard errors, adjusting for the baseline score as a precision variable; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-0.8 to 3.2]

7. Secondary Outcome: Number of Participants Reporting Suicide Attempts as Measured by the Columbia Suicide Severity Rating Scale & Completed Suicide
Description: Three elements of the full version of the Columbia Suicide Severity Rating Scale (C-SSRS) (lifetime-recent (baseline) and since last visit (6 months)) were complied to create a Suicide Attempts Survey. These measured self-reported aborted or self-interrupted suicide attempts, interrupted suicide attempts, and actual suicide attempts. Non-lethal self-harm and lethal means used for attempts or completions were also collected. These elements were not included in the C-SSRS score but were compared across the intervention groups. Medical records were used to measure suicide completion.
Time Frame: Baseline and 6 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Patients - CC | Patients - CC+ | Healthcare Providers/Staff - CC | Healthcare Providers/Staff - CC+
Number analyzed (Participants) | 166 | 165 | 168 | 167
Participants
  Death by suicide | 0 | 0 | 1 | 0
  Attempted suicide | 0 | 0 | 2 | 0
  Interrupted/aborted suicide | 0 | 1 | 3 | 3

8. Secondary Outcome: Number of Participants Reporting Increased Alcohol, Tobacco, Marijuana, and Illicit Drug Use as Measured by Questions Adapted From Youth Risk Behavior Survey and Related to COVID-19
Description: The questions are adapted from the Youth Risk Behavior Survey and will contain additional questions to measure self-reported changes in alcohol or illicit-drug use since the beginning of the COVID-19 pandemic.
Time Frame: Baseline and 6 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Patients - CC | Patients - CC+ | Healthcare Providers/Staff - CC | Healthcare Providers/Staff - CC+
Number analyzed (Participants) | 166 | 165 | 168 | 167
Participants
  Increased tobacco use at follow-up (6 months): number analyzed (Participants) | 163 | 152 | 164 | 164
  Increased tobacco use at follow-up (6 months) | 23 | 13 | 16 | 6
  Increased alcohol use at follow-up (6 months): number analyzed (Participants) | 162 | 153 | 164 | 162
  Increased alcohol use at follow-up (6 months) | 42 | 38 | 52 | 55
  Increased marijuana/cannabis use at follow-up (6 months): number analyzed (Participants) | 156 | 152 | 156 | 159
  Increased marijuana/cannabis use at follow-up (6 months) | 15 | 19 | 17 | 14
  Increased illicit drug use at follow-up (6 months): number analyzed (Participants) | 159 | 157 | 159 | 165
  Increased illicit drug use at follow-up (6 months) | 7 | 3 | 3 | 2
Statistical Analysis 1: Comparison: Patients - CC vs Patients - CC+; Number of participants with increased tobacco use among patients randomized to CC+ vs CC; Test type: Superiority; p = 0.12, GLM — p<0.05 = a priori threshold for statistical significance; Generalized linear model (GLM) with an identity link and binomial variance; Risk Difference (RD) = -5.6, 95% CI 2-sided [-12.5 to 1.4]
Statistical Analysis 2: Comparison: Healthcare Providers/Staff - CC vs Healthcare Providers/Staff - CC+; Number of participants with increased tobacco use among healthcare providers/staff randomized to CC+ vs CC; Test type: Superiority; p = 0.03, GLM — p<0.05 = a priori threshold for statistical significance; Generalized linear model (GLM) with an identity link and binomial variance; Risk Difference (RD) = -6.1, 95% CI 2-sided [-11.5 to -0.7]
Statistical Analysis 3: Comparison: Patients - CC vs Patients - CC+; Number of participants with increased alcohol use among patients randomized to CC+ vs CC; Test type: Superiority; p = 0.83, GLM — p<0.05 = a priori threshold for statistical significance; Generalized linear model (GLM) with an identity link and binomial variance; Risk Difference (RD) = -1.1, 95% CI 2-sided [-10.7 to 8.5]
Statistical Analysis 4: Comparison: Healthcare Providers/Staff - CC vs Healthcare Providers/Staff - CC+; Number of participants with increased alcohol use among healthcare providers/staff randomized to CC+ vs CC; Test type: Superiority; p = 0.67, GLM — p<0.05 = a priori threshold for statistical significance; Generalized linear model (GLM) with an identity link and binomial variance; Risk Difference (RD) = 2.2, 95% CI 2-sided [-8.0 to 12.5]
Statistical Analysis 5: Comparison: Patients - CC vs Patients - CC+; Number of participants with increased marijuana/cannabis use among patients randomized to CC+ vs CC; Test type: Superiority; p = 0.42, GLM — p<0.05 = a priori threshold for statistical significance; Generalized linear model (GLM) with an identity link and binomial variance; Risk Difference (RD) = 2.9, 95% CI 2-sided [-4.1 to 9.9]
Statistical Analysis 6: Comparison: Healthcare Providers/Staff - CC vs Healthcare Providers/Staff - CC+; Number of participants with increased marijuana/cannabis use among healthcare providers/staff randomized to CC+ vs CC; Test type: Superiority; p = 0.53, GLM — p<0.05 = a priori threshold for statistical significance; Generalized linear model (GLM) with an identity link and binomial variance; Risk Difference (RD) = -2.1, 95% CI 2-sided [-8.7 to 4.5]
Statistical Analysis 7: Comparison: Patients - CC vs Patients - CC+; Number of participants with increased illicit drug use among patients randomized to CC+ vs CC; Test type: Superiority; p = 0.20, GLM — p<0.05 = a priori threshold for statistical significance; Generalized linear model (GLM) with an identity link and binomial variance; Risk Difference (RD) = -2.5, 95% CI 2-sided [-6.3 to 1.4]
Statistical Analysis 8: Comparison: Healthcare Providers/Staff - CC vs Healthcare Providers/Staff - CC+; Number of participants with increased illicit drug use among healthcare providers/staff randomized to CC+ vs CC; Test type: Superiority; p = 0.62, GLM — p<0.05 = a priori threshold for statistical significance; Generalized linear model (GLM) with an identity link and binomial variance; Risk Difference (RD) = -0.7, 95% CI 2-sided [-3.4 to 2.0]

9. Secondary Outcome: Number of Participants Who Attended Mental Healthcare Appointments: Self-Report
Description: Participant engagement in outpatient mental health services will be measured as a dichotomous variable through self-report.
Time Frame: 6 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Patients - CC | Patients - CC+ | Healthcare Providers/Staff - CC | Healthcare Providers/Staff - CC+
Number analyzed (Participants) | 166 | 165 | 168 | 167
Participants | 119 | 105 | 124 | 123
Statistical Analysis 1: Comparison: Patients - CC vs Patients - CC+; Difference in proportion of patients attending mental healthcare appointments by intervention arm at follow-up (6 months); Test type: Superiority; p = 0.41, GLM — p<0.05 = a priori threshold for statistical significance; Generalized linear model (GLM) with an identity link and binomial variance; Risk Difference (RD) = -4.5, 95% CI 2-sided [-15.4 to 6.3]
Statistical Analysis 2: Comparison: Healthcare Providers/Staff - CC vs Healthcare Providers/Staff - CC+; Difference in proportion of healthcare providers/staff attending mental healthcare appointments by intervention arm at follow-up (6 months); Test type: Superiority; p = 0.31, GLM — p<0.05 = a priori threshold for statistical significance; Generalized linear model (GLM) with an identity link and binomial variance; Risk Difference (RD) = 5.5, 95% CI 2-sided [-5.2 to 16.2]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Patients - CC | Patients - CC+ | Healthcare Providers/Staff - CC | Healthcare Providers/Staff - CC+
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/165 | 1/168 | 0/167
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/165 | 0/168 | 0/167
Other Adverse Events (participants affected / at risk) | 0/166 | 0/165 | 0/168 | 0/167

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-12-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT04700137/Prot_001.pdf
  • Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT04700137/SAP_002.pdf
  • Informed Consent Form (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT04700137/ICF_000.pdf